CLINICAL TRIAL: NCT07025980
Title: Effect of Sinbiotic With Multispecies Probiotics on Liver Parameters in Patients With Metabolic Associated Steatotic Liver Disease
Brief Title: Effect of Sinbiotic With Multispecies Probiotics on Liver Parameters Liver Enzymes, Ultrasound, Elastography and Adipokines in Same Cases) in Patients With Metabolic Associated Steatotic Liver Disease.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eva Cubric (Other)
Collaborators: General Hospital Šibenik, Croatia (Other); General Hospital Zadar (Other); University Hospital Dubrava (Other); University Hospital Rijeka (Other); Clinical Hospital Merkur (Other); University Hospital Sestre Milosrdnice (Other); University Hospital of Split (Other)
Responsible Party: Sponsor-Investigator, Eva Cubric, doctor medicine, General Hospital Šibenik, Croatia
Organization: General Hospital Šibenik, Croatia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-22682/1-23
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: MASLD/MASH (Metabolic Dysfunction-Associated Steatotic Liver Disease / Metabolic Dysfunction-Associated Steatohepatitis); Diabetes Mellitus; Hypertension; Hyperlipidaemia
Keywords: elastography; human LRG1, liver enzymes, metabolic- dysfuncion steatotic liver disease, metabolic syndrome; probiotics, treatment
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: This is a randomized, multicenter, double-blind clinical trial. If they meet the inclusion criteria at the next medical examination (study start-randomization period) upon entering the study, patients will be randomized into two groups in a 1:1 ratio, where one group will receive the test product (n=57) and the other/control group placebo (n=57).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test group (Experimental): Test group (n 57) The test product is a ready-to-use preparation PROBalansHepatocare, manufactured by PharmaS d.o.o., which contains 8 strains of live cultures of microorganisms (Bifidobacteriumbreve BBR8, Bifidobacteriuminfantis SP37, Bifidobacteriumlongum SP54, Lactobacillus acidophilus LA1, Lactobacillus bulgaricus LB2, Lactobacillus paracasei IMC502®, Lactobacillus plantarum BG 112, Streptococcusthermophilus SP4) with about 100 billion bacteria (50x109 CFU/capsule) in two capsules per day. In addition, the test product contains 100 mg of fructooligosaccharides, 210 mg of Ca-butyrate, and 10 ug (400 IU) of vitamin D in each capsule.
  Interventions: Dietary Supplement: The test product is a ready-to-use sinbiotic preparation of multispecies probiotics, ca-butyrate and FOS
- Placebo (Placebo Comparator): Placebo group (n 57)The placebo is identical to the test product in all aspects (organoleptic), but contains only excipients (cellulose; hydroxypropyl-methyl cellulose) and 10 ug (400 IU) of vitamin D.
  Interventions: Dietary Supplement: Placebo Drug

INTERVENTIONS:
Dietary Supplement: The test product is a ready-to-use sinbiotic preparation of multispecies probiotics, ca-butyrate and FOS — The test product is a ready-to-use preparation PROBalansHepatocare, manufactured by PharmaS d.o.o., which contains 8 strains of live cultures of microorganisms (Bifidobacteriumbreve BBR8, Bifidobacteriuminfantis SP37, Bifidobacteriumlongum SP54, Lactobacillus acidophilus LA1, Lactobacillus bulgaricus LB2, Lactobacillus paracasei IMC502®, Lactobacillus plantarum BG 112, Streptococcusthermophilus SP4) with about 100 billion bacteria (50x109 CFU/capsule) in two capsules per day. In addition, the test product contains 100 mg of fructooligosaccharides, 210 mg of Ca-butyrate, and 10 ug (400 IU) of vitamin D in each capsule.
  Arms: test group
Dietary Supplement: Placebo Drug — Contains only excipients (cellulose; hydroxypropyl-methyl cellulose) and 10 ug (400 IU) of vitamin D. They do not contain dyes, flavors or preservatives, and contain traces of soy and milk, the levels of which do not affect people who are lactose intolerant.
  Arms: Placebo

SUMMARY:
Scientific hypothesis: the use of a synbiotic preparation with a multi-strain probiotic in patients with MASLD can lead to a decrease in non-invasive elastographic parameters of hepatic steatosis and fibrosis and an improvement in liver function.

The main objective of this study is to examine whether the test product affects the improvement of liver function measured by elastographic parameters or at least the prevention of further disease progression.

The goal of this clinical trial is to learn if sinbiotics works to improve liver function in adult patients with MASLD The main questions it aims to answer are:

Does sinbiotic lowers elastographic parameters od steatosis and fibrosis? Does it change liver function by lowering liver enzymes, blood lipids and sugar? Can sinbiotics lower CV risks and improve quality of life? Researchers will compare sinbiotic to a placebo (a look-alike substance that contains no drug) to see if sinbiotic works in MASLD patients.

Participants will:

Take sinbiotic or a placebo every day (td) for 9 months Visit the clinic once every 3 months for checkups, and at the begining and after 9 months for blood tests and US with elastography Keep a diary of their symptoms, diet, activity

DETAILED DESCRIPTION:
This is a randomized, multicenter, double-blind 1:1 clinical study lasting 3 years, which is planned to begin on January 2, 2025. The study will include 114 patients of both sexes over the age of 18, who suffer from MASLD and are monitored in the gastroenterology and/or endocrinology outpatient department of the Šibenik-Knin County General Hospital and cooperating institutions (Sestara milosrdnica Clinical Hospital, Split Clinical Hospital, Dubrava Clinical Hospital, Merkur Clinical Hospital, Požega General and County Hospital, Zadar General Hospital, Rijeka Clinical Hospital). Patients will take the prepared preparation (synbiotic or placebo) for 36 weeks at a dose of 2x1 capsule per day. During the study, they will keep a diary of consumption and possible side effects, and every three months they will pick up coded packages of the preparation at the gastroenterology clinic of their institution. Cooperation will be checked by telephone calls and by reviewing the diary at monthly intervals, and more often if necessary. Patients will regularly take their usual chronic therapy, especially antihypertensives, antidiabetics, and hypolipidemics, they will be recommended appropriate physical activity during the week and a diet in accordance with the recommendations of professional societies, and the use of herbal preparations and other dietary supplements is prohibited. Serum samples will be taken from the patients at the beginning of the study and at the end of the intervention for routine biochemical tests, and for the ELISA test of human LRG1 and adiponectin in some centers (after 9 months of using the test preparation or placebo). In addition to the above, an ultrasound of the liver, Fibrocan, and in some centers elastography on an Aloka Arietta ultrasound system will be performed in the same interval. All patients will have their BMI, waist circumference, and arterial pressure values measured using a standard method, and they will complete a questionnaire on quality of life and the SCORE2 CV risk table.

ELIGIBILITY:
Inclusion Criteria:

* MASLD confirmed by ultrasound and elastography with CAP > 260 dB/m/MHz;
* other causes of chronic liver disease excluded and/or diagnosis confirmed by liver biopsy,
* presence of metabolic syndrome according to the definition of the International Diabetes Federation (IDF): waist circumference for women over 80 cm or over 94 cm for men, and at least two of the other criteria (treated hypertensive or blood pressure > 130/85 mmHg determined during inclusion; treated diabetic or newly detected fasting serum glucose levels > 5.6 mmol/l; treated dyslipidemia or newly detected serum triglyceride levels > 1.7 mmol/L or HDL < 1.29 mmol/L for women/< 1.03 mmol/L for men),
* signed informed consent.

Exclusion Criteria:

* pregnancy,
* significant alcohol intake (>30g/day in men, >20g/day in women),
* presence of autoimmune, viral, cholestatic (primary biliary cholangitis, primary sclerosing cholangitis, obstructive biliary tree diseases) or metabolic (hemochromatosis, Wilson) causes of chronic liver disease, transplant patients, malignant diseases, free fluid in the abdomen, significant small bowel resections,
* signs of liver cirrhosis or LSM>13 kPa measured TE,
* use of medications that can promote the development of steatosis (e.g. corticosteroids, high doses of estrogen, methotrexate, amiodarone, valproate), and medications that can affect the composition of the microbiota for at least 3 months before the start of the study (antibiotics and probiotics),
* inability to reliably measure CAP and LSM (IQR/median>30%),
* severe psychiatric patients in whom cooperation and consent are questionable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
change in the controlled attenuated coefficient CAP (dB/m/MHZ) for steatosis | at baseline and after 270 days of intervention*
change in liver stiffness measurement (LSM) (kPa) measured by transient elastography for fibrosis | at baseline and after 270 days of intervention
  (1st and 2nd measured on FibroScan device, manufacturer Echosens, Paris, France)

SECONDARY OUTCOMES:
change in serum levels of aspartate aminotransferase AST (U/L), alanine transferase ALT (U/L), gamma-glutamyl transferase GGT (U/L), ferritin (ng/ml) | at baseline and after 270 days
change in serum levels of glucose (mmol/l) and fasting insulin (pmol/L), calculation of insulin resistance using the Homeostatic Model Assessment for Insulin Resistance formula HOMA-IR (glucose (mmol/l) x insulin (pmol/L)/22.5) | at baseline and after 270 days
change in serum levels of cholesterol (mmol/L), triglycerides (mmol/L), HDL-cholesterol (mmol/L) and LDL-cholesterol (mmol/L) | at baseline and after 270 days
change in waist circumference (cm) and body mass index (BMI=body weight (kg)/body height2(m)), kg/m2) | at baseline and after 270 days
change in blood pressure (mmHg) measured by standard method | at baseline and after 270 days
change in human Leucin-rich alpha-2-gylcoprotein 1 (LRG1) (ng/ml) | at baseline and after 270 days
  ELISA test BIOSOURCE
change in fecal calprotectin (ug/g) | at baseline and after 270 days
change in controlled attenuated coefficient ATT (dB/cm/MHZ) for steatosis | at baseline and after 270 days of intervention*
change in liver stiffness (Elastography) E (kPa) measured by 2D SWE for fibrosis | at baseline and after 270 days of intervention
  ATT and E measured on Aloka Arrieta US system, by FUJI; Tokyo, Japan
change in cardiovascular risk according to the European Society of Cardiology SCORE-2 tables | at baseline and after 270 days
  SCORE-2 tables for high risk population
change in quality of life according to the validated WHO SF-36 Quality of Life Questionnaire | at baseline and after 270 days
change in serum adiponectin levels (ng/ml) | at baseline and after 270 days (only on Sibenik patients)
  ELISA human test, Biosource

CONTACTS AND LOCATIONS:
Overall Officials: Marko Skelin, ass.prof.dr.sc, mag.pharm., Study Chair — GH Sibenik-Knin County, Medical Faculty University of Rijeka, Croatia
Locations (1):
- General Hospital Sibenik-Knin County, Šibenik, Croatia, Croatia

IPD SHARING:
Plan to Share IPD: No
It will not be shared in public, but by the individual request, and only after the approval of each institution in collaboration (as Ethics Commities of each institution has demand)

REFERENCES:
- [Background] Lukenda Zanko V, Domislovic V, Trkulja V, Krznaric-Zrnic I, Turk-Wensveen T, Krznaric Z, Filipec Kanizaj T, Radic-Kristo D, Bilic-Zulle L, Orlic L, Dinjar-Kujundzic P, Poropat G, Stimac D, Hauser G, Mikolasevic I. Vitamin D for treatment of non-alcoholic fatty liver disease detected by transient elastography: A randomized, double-blind, placebo-controlled trial. Diabetes Obes Metab. 2020 Nov;22(11):2097-2106. doi: 10.1111/dom.14129. Epub 2020 Aug 5. PMID 32613718
- [Background] Fogacci F, Giovannini M, Di Micoli V, Grandi E, Borghi C, Cicero AFG. Effect of Supplementation of a Butyrate-Based Formula in Individuals with Liver Steatosis and Metabolic Syndrome: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Nutrients. 2024 Jul 28;16(15):2454. doi: 10.3390/nu16152454. PMID 39125336
- [Background] Silva RSD, Mendonca IP, Paiva IHR, Souza JRB, Peixoto CA. Fructooligosaccharides and galactooligosaccharides improve hepatic steatosis via gut microbiota-brain axis modulation. Int J Food Sci Nutr. 2023 Nov;74(7):760-780. doi: 10.1080/09637486.2023.2262779. Epub 2023 Nov 15. PMID 37771001
- [Background] Duseja A, Acharya SK, Mehta M, Chhabra S; Shalimar; Rana S, Das A, Dattagupta S, Dhiman RK, Chawla YK. High potency multistrain probiotic improves liver histology in non-alcoholic fatty liver disease (NAFLD): a randomised, double-blind, proof of concept study. BMJ Open Gastroenterol. 2019 Aug 7;6(1):e000315. doi: 10.1136/bmjgast-2019-000315. eCollection 2019. PMID 31423319
- [Background] Dong TS, Jacobs JP. Nonalcoholic fatty liver disease and the gut microbiome: Are bacteria responsible for fatty liver? Exp Biol Med (Maywood). 2019 Apr;244(6):408-418. doi: 10.1177/1535370219836739. Epub 2019 Mar 14. PMID 30871368
- [Background] Khan A, Ding Z, Ishaq M, Bacha AS, Khan I, Hanif A, Li W, Guo X. Understanding the Effects of Gut Microbiota Dysbiosis on Nonalcoholic Fatty Liver Disease and the Possible Probiotics Role: Recent Updates. Int J Biol Sci. 2021 Feb 8;17(3):818-833. doi: 10.7150/ijbs.56214. eCollection 2021. PMID 33767591
- [Background] Bozic D, Podrug K, Mikolasevic I, Grgurevic I. Ultrasound Methods for the Assessment of Liver Steatosis: A Critical Appraisal. Diagnostics (Basel). 2022 Sep 22;12(10):2287. doi: 10.3390/diagnostics12102287. PMID 36291976
- [Background] Merriman RB, Ferrell LD, Patti MG, Weston SR, Pabst MS, Aouizerat BE, Bass NM. Correlation of paired liver biopsies in morbidly obese patients with suspected nonalcoholic fatty liver disease. Hepatology. 2006 Oct;44(4):874-80. doi: 10.1002/hep.21346. PMID 17006934
- [Background] Sanyal AJ, Williams SA, Lavine JE, Neuschwander-Tetri BA, Alexander L, Ostroff R, Biegel H, Kowdley KV, Chalasani N, Dasarathy S, Diehl AM, Loomba R, Hameed B, Behling C, Kleiner DE, Karpen SJ, Williams J, Jia Y, Yates KP, Tonascia J. Defining the serum proteomic signature of hepatic steatosis, inflammation, ballooning and fibrosis in non-alcoholic fatty liver disease. J Hepatol. 2023 Apr;78(4):693-703. doi: 10.1016/j.jhep.2022.11.029. Epub 2022 Dec 14. PMID 36528237
- [Background] Buzzetti E, Pinzani M, Tsochatzis EA. The multiple-hit pathogenesis of non-alcoholic fatty liver disease (NAFLD). Metabolism. 2016 Aug;65(8):1038-48. doi: 10.1016/j.metabol.2015.12.012. Epub 2016 Jan 4. PMID 26823198
- [Background] Kobyliak N, Abenavoli L, Mykhalchyshyn G, Kononenko L, Boccuto L, Kyriienko D, Dynnyk O. A Multi-strain Probiotic Reduces the Fatty Liver Index, Cytokines and Aminotransferase levels in NAFLD Patients: Evidence from a Randomized Clinical Trial. J Gastrointestin Liver Dis. 2018 Mar;27(1):41-49. doi: 10.15403/jgld.2014.1121.271.kby. PMID 29557414
- [Background] Rinella ME, Neuschwander-Tetri BA, Siddiqui MS, Abdelmalek MF, Caldwell S, Barb D, Kleiner DE, Loomba R. AASLD Practice Guidance on the clinical assessment and management of nonalcoholic fatty liver disease. Hepatology. 2023 May 1;77(5):1797-1835. doi: 10.1097/HEP.0000000000000323. Epub 2023 Mar 17. No abstract available. PMID 36727674